CLINICAL TRIAL: NCT06656572
Title: Immunogenomic Analyses of Pediatric Catatonia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rady Pediatric Genomics & Systems Medicine Institute (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Aaron Besterman, Health Sciences Associate Clinical Professor, UCSD Department of Psychiatry Clinical Investigator, Rady Children's Institute for Genomic Medicine Child & Adolescent Psychiatrist, Rady Children's Hospital San Diego, Rady Pediatric Genomics & Systems Medicine Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 810014; 314882-00001 (Other Grant/Funding Number: Brain and Behavior Research Foundation)
Record Dates: First submitted 2024-10-22; First posted 2024-10-24 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Catatonia
Keywords: Genomics; Pediatric
MeSH Terms: conditions — Catatonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Enrollees - WGS (Experimental): These participants will be subject to whole genome sequencing and Phage ImmunoPrecipiation sequencing (PhIP-Seq) to identify genetic changes and novel antibodies associated with catatonia.
  Interventions: Genetic: Genetic: Genomic sequencing and molecular diagnostic results, if any.; Diagnostic Test: Phage display ImmunoPrecipiation Sequencing (PhIP-Seq)

INTERVENTIONS:
Genetic: Genetic: Genomic sequencing and molecular diagnostic results, if any. — Genomic sequencing results may be used for diagnosis and treatment of participants.
Diagnostic Test: Phage display ImmunoPrecipiation Sequencing (PhIP-Seq) — Whole Proteome programmable phage display immunoprecipitation sequencing will be used to diagnose known and novel autoantibodies.

SUMMARY:
Rady Children's Institute for Genomic Medicine seeks to understand the genomes and immune systems in 40 children and adolescents who are admitted to Rady Children's Hospital San Diego with a catatonia diagnosis. Cutting-edge genome and protein sequencing technology will be used to better understand how immunological and genetic assessments may improve the ability to identify the cause of catatonia and impact care. The investigator also hopes to identify new genetic and/or autoimmune causes of catatonia that may inform new treatment for future patients.

DETAILED DESCRIPTION:
Catatonia is a complex condition that affects children's behavior, movement, and emotions. It can be caused by various underlying health issues, such as genetic disorders or problems with the immune system. Identifying these underlying causes is crucial for providing the best care and treatment to affected children. In this study, the investigators aim to compare the effectiveness of traditional medical tests with a more advanced approach that includes genetic testing and immune system screening in finding the underlying causes of catatonia in children. The investigators will compare two groups of children with catatonia. One group will be identified from hospital records and will have undergone standard medical tests to find the cause of their catatonia. The other group will be a new set of patients who will receive both standard medical tests and additional advanced testing, including genome sequencing (a technique that reads the entire genetic code) and screening for antibodies that attack the brain. The investigators will use a statistical method called propensity score matching to make sure that the two groups are as similar as possible in terms of age, sex, and other relevant factors. This will help the investigators to fairly compare the effectiveness of the two approaches in identifying the underlying causes of catatonia. The investigators expect that combining standard medical tests with genome sequencing and autoantibody screening will be more effective in finding the underlying causes of catatonia in children compared to using standard medical tests alone. This could lead to more accurate diagnoses and more targeted treatments for children with catatonia, helping them to recover more quickly and improving their quality of life. If this study shows that the advanced testing approach is more effective in finding the underlying causes of catatonia, this could change the way doctors approach the diagnosis and treatment of this complex condition. In turn, this could lead to more accurate diagnoses, tailored treatments, and improved outcomes for children with catatonia and their families.

ELIGIBILITY:
Inclusion Criteria:

* Individual in whom one of the following criteria is met:

  1. Child/adolescent Ages 0-17 (2) with a diagnosis of catatonia.

     OR
  2. Biological parents of child/adolescent enrolled in this study for the purposes of reflex testing. Family members are eligible for participation in this study if they are presumed to be genetically related to a patient participant

Exclusion Criteria:

* Child/adolescents patients who do not meet any of the inclusion criteria, or those who:

  1. Already received any prior whole genome sequencing or exome sequencing.
  2. Unable to approach the family or patient for enrollment.
  3. Unable to obtain informed consent.
  4. Family members are ineligible for participation in this study if:

     1. They are known to not be genetically related to the child/adolescent patient participant

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic rate of whole genome sequencing | 2 years
  Evaluate the impact of whole genome sequencing on diagnostic yield in pediatric catatonia, compared to standard medical workup.
Diagnostic rate of brain reactive autoantibodies | 2 years
  Diagnostic rate of brain reactive autoantibodies via genomic and whole human proteome programmable phage display immunoprecipitation sequencing (PhIP-Seq)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Besterman, MD, Principal Investigator — Rady Pediatric Genomics & Systems Medicine Institute